CLINICAL TRIAL: NCT00494208
Title: Testosterone Dose Response in Surgically Menopausal Women
Brief Title: TDSM- Testosterone Dose Response in Surgically Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U54HD041748 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2009-01

CONDITIONS: Hysterectomy; Ovariectomy; Menopause; Testosterone Deficiency
Keywords: androgens; testosterone; testosterone deficiency; women; menopause; surgical Menopause; hysterectomy; oophorectomy; ovariectomy; sexual dysfunction; sexual function; muscle function; insulin sensitivity; body composition
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Insulin Resistance | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- 1 (Active Comparator)
  Interventions: Drug: Testosterone
- 2 (Active Comparator)
  Interventions: Drug: Testosterone
- 3 (Active Comparator)
  Interventions: Drug: Testosterone
- 4 (Active Comparator)
  Interventions: Drug: Testosterone
- 5 (Active Comparator)
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Testosterone ester

SUMMARY:
TDSM will study the physiology of testosterone in women ages 21-60 who have had surgical menopause (uterus and both ovaries removed). Testosterone is commonly thought of as a "male hormone" thus being that it is the male's primary hormone. Women produce testosterone in much smaller amounts and despite this, testosterone still plays a significant role. Fifty percent of a women's testosterone is made in her adrenal glands (glands that sit on top of the kidneys) and fifty percent is made in her ovaries. When a woman has her ovaries removed it is thought that her testosterone levels decrease rapidly and significantly. This study will be examining testosterone's role in sexual function, general well being, muscle performance, cognitive function, carbohydrate metabolism and muscle and fat distribution.

The study is 14 months long with weekly to monthly visits. The subjects will be placed on the estrogen patch for the duration of the study. They will also be given weekly injections of testosterone or placebo for 6 months. During the testosterone treatment phase the women will be separated into 5 groups. The groups include a dose of testosterone that is very low, low, medium, high and placebo. A placebo looks and feels similar to testosterone; however it does not have testosterone in it. We use this to test if the subject is having a response to the testosterone itself or the thought of receiving testosterone. Neither the subject nor the investigators will know the dose until the end of the study.

DETAILED DESCRIPTION:
In healthy women the primary hormones produced by the ovaries are estrogens and progesterone, but they also produce testosterone both before and after menopause. Although normal blood levels of testosterone in women are much lower than in men, testosterone is thought to have important physiologic effects in women, particularly on muscle function, body composition, sexual function and cognitive function. When women require bilateral oophorectomy (removal of ovaries), they subsequently have a significant drop in serum testosterone levels. They also frequently experience a decreased sense of well being, and decreased sexual function.

While treatment with testosterone and other androgens has been widely promoted for women with low serum levels, there is little available data on the effects of such treatment particularly when given in physiologic doses (doses resulting in normal blood levels for women). Studies that have demonstrated benefits of testosterone in women have often used doses of testosterone which resulted in higher than normal serum testosterone levels. At such doses, testosterone and other androgens can produce virilizing side effects such as increased facial and body hair, acne, increased size of the clitoris and changes in the voice.

It is not known whether physiologic testosterone replacement can provide the benefits seen with higher doses in women with androgen deficiency without the limiting, virilizing side effects. It has been assumed that testosterone dose-response relationships are different in women than in men, and that clinically significant effects on psycho-sexual function, body composition, muscle performance, cognitive function, and other health-related outcomes can be achieved at testosterone doses and concentrations that are substantially lower than those required to produce similar effects in men; however, these assumptions have not been tested rigorously.

Therefore, the primary objective of this study is to establish testosterone dose-response relationships in surgically menopausal women with low testosterone concentrations for a range of androgen-dependent outcomes, including sexual function, fat-free mass, thigh muscle strength and leg power, several domains of neurocognitive function, plasma lipids, apolipoproteins and lipoprotein particles, and insulin sensitivity.

The secondary objective is to determine the range of testosterone doses and subsequent plasma testosterone concentrations that are associated with improvements in sexual, physical and neurocognitive functions and that can be safely administered to women without significant adverse effects on hair growth, voice, sebum production, clitoral size, and cardiovascular risk factors.

Hypotheses

1. Testosterone administration in surgically menopausal women with low testosterone concentrations is associated with dose- and concentration-dependent improvements in sexual function and sexual activity scores, specific domains of cognitive function, fat-free mass, thigh muscle strength, and leg power.
2. Testosterone dose-response relationships are different for different androgen dependent processes. While some domains of sexual function are normalized by testosterone concentrations at the upper end of the normal range for healthy, young women, significant gains in fat-free mass, thigh muscle strength and power would require higher testosterone doses than those required to induce changes in sexual function.

ELIGIBILITY:
Inclusion Criteria

* Medically stable, ambulatory, surgically menopausal women, 21-60 years of age, who have undergone bilateral salpingo-oophorectomy and hysterectomy at least 6 months before study entry
* Serum total testosterone concentrations less than 31 ng/dL or free testosterone less than 3.5 pg/ml (less than the median for healthy, young women
* Able to understand and give informed consent.
* The women will have been on a stable regimen of transdermal estrogen replacement for at least three months. Those who are not on estrogen replacement or are taking a different mode of estrogen replacement will be included only if they are willing to switch to transdermal estradiol patch (see below).
* A normal PAP smear (if subject has a cervix) and mammogram in the preceding 12 months.

Exclusion Criteria:

* Significant depression, as assessed by Beck's Depression Scale.
* Any acute or chronic illness, malignant disease or fever of known or unknown origin will be excluded.
* Poorly controlled diabetes mellitus (hemoglobin A1c greater than 8.5%)
* Uncontrolled hypertension defined as blood pressure of greater than 160/100
* Severe obesity defined as body mass index of greater than 40 kg/m2
* Current or recent (last 6 months) users of illicit drugs (which may affect appetite, food intake, metabolism, and/or compliance with the protocol)
* Any one planning to initiate a weight-reduction diet in the subsequent six months
* Alcohol or drug dependence currently or in the preceding 6 month.
* Significant liver function abnormalities, defined as SGOT, SGPT or alkaline phosphatase value of greater than three times the upper limit of normal in our Clinical Pathology Laboratory or serum bilirubin levels of greater than 1.5 mg/dl will be excluded.
* History of breast, ovarian, endometrial or cervical cancer
* History of hyperandrogenic disorders such as hirsutism, grade 2 or 3 acne, and polycystic ovary disease. Testosterone administration to these patients may exacerbate the underlying disorder.
* Intolerance to other transdermal formulations
* Women with abnormal PAP smears or mammograms will not be included unless they have been evaluated by their gynecologists and breast and uterine/cervical cancers have been excluded by appropriate tests.
* Women with dementia as assessed by the mini-mental state examination
* Women with depression, assessed by Beck's Depression Scale.
* Those with disabilities that would prevent them from participating in strength testing (e.g., amputation of limbs, blindness, severe arthritis, neurologic disorders such as Parkinson's disease, stroke, or myopathy).
* Women with any heart disease, including angina, congestive heart failure, or history of myocardial infarction or coronary artery angioplasty or bypass surgery in the previous year will be excluded.
* Subjects planning to initiate a weight-reduction diet in the subsequent six months
* Other Medications. Women who have received in the preceding three months drugs known to affect testosterone production or metabolism such as ketoconazole, Megace, and/or anabolic/androgenic steroids will be excluded. We will also exclude women who are taking or have taken in the past three months medication that include sexual dysfunction (e.g., spironolactone, SSRIs, GnRH agonists). Women who are using any medication, device or dietary supplement known to enhance sexual function will not be included. Women receiving thyroid hormone replacement therapy may participate in the study only if they have been on a stable replacement dose of L-thyroxine for at least three months.
* Intolerance to estrogen products or skin patches
* Undiagnosed vaginal or vulvar bleeding
* History of deep vein thrombosis, pulmonary embolism, or other thromboembolic disorder

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Physical Function | 14 months

SECONDARY OUTCOMES:
Muscle mass | 14 months
Lipids, glucose, HOMA | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Boston Univeristy Medical Center; Shehzad Basaria, M.D., Study Director — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Tapper J, Huang G, Pencina KM, Li Z, Arver S, Martling A, Blomqvist L, Buchli C, Travison TG, Storer TW, Bhasin S, Basaria S. The effects of testosterone administration on muscle areas of the trunk and pelvic floor in hysterectomized women with low testosterone levels: proof-of-concept study. Menopause. 2019 Dec;26(12):1405-1414. doi: 10.1097/GME.0000000000001410. PMID 31479032
- [Derived] Huang G, Pencina KM, Coady JA, Beleva YM, Bhasin S, Basaria S. Functional Voice Testing Detects Early Changes in Vocal Pitch in Women During Testosterone Administration. J Clin Endocrinol Metab. 2015 Jun;100(6):2254-60. doi: 10.1210/jc.2015-1669. Epub 2015 Apr 15. PMID 25875779
- [Derived] Huang G, Tang E, Aakil A, Anderson S, Jara H, Davda M, Stroh H, Travison TG, Bhasin S, Basaria S. Testosterone dose-response relationships with cardiovascular risk markers in androgen-deficient women: a randomized, placebo-controlled trial. J Clin Endocrinol Metab. 2014 Jul;99(7):E1287-93. doi: 10.1210/jc.2013-4160. Epub 2014 Apr 8. PMID 24712568
- [Derived] Huang G, Basaria S, Travison TG, Ho MH, Davda M, Mazer NA, Miciek R, Knapp PE, Zhang A, Collins L, Ursino M, Appleman E, Dzekov C, Stroh H, Ouellette M, Rundell T, Baby M, Bhatia NN, Khorram O, Friedman T, Storer TW, Bhasin S. Testosterone dose-response relationships in hysterectomized women with or without oophorectomy: effects on sexual function, body composition, muscle performance and physical function in a randomized trial. Menopause. 2014 Jun;21(6):612-23. doi: 10.1097/GME.0000000000000093. PMID 24281237